CLINICAL TRIAL: NCT06805929
Title: Correlation Study Between Clinical, Neurophysiological, and Neuroradiological Biomarkers and Rehabilitation Outcomes to Predict Functional Recovery After Stroke and Personalize Treatment.
Brief Title: Correlation Between Clinical Neurological Biomarkers and Rehabilitation Outcome
Acronym: PREVICTUS
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 20/15
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our study purpose is to evaluate the predictive power of various clinical, neurophysiological, and neuroimaging biomarkers-acquired and analyzed using advanced and integrated techniques-on motor functional recovery and disability post-stroke. The goal is to construct an integrated individual biomarker algorithm with a high predictive value for outcomes.

DETAILED DESCRIPTION:
Ability to predict post-stroke individual recovery still represents an important challenge to develop personalized and effective neurorehabilitation strategies. The aim of this study is to verify the predictive power of different clinical, neurophysiological and neuroimaging biomarkers in combination, acquired and analysed using advanced, integrated techniques, on functional motor recovery and post-stroke disability.

Patients with ischemic or hemorrhagic stroke and hemiparesis are subsequently enrolled and undergo multimodal assessment that includes measures spanning 4 assessment categories: demographic/medical history, clinical biomarkers, neurophysiological biomarkers (Motor Evoked Potentials, High-density EEG), neuroimaging biomarkers (infarct volume, corticospinal tract injury) at T0 (from 14 to 30 days post-stroke), T1 (after 2 months of intensive rehabilitation treatment) and T2 (4-6 months after discharge). Primary endpoint is change in arm Fugl-Meyer score. Secondary endpoints are changes in lower limb Fugl Meyer motor, Nine hole peg test, National Institute of Health Stroke Scale, mRS Rankin Scale, modified Barthel Index scores.

Multivariate analyses will indicate which biomarkers at baseline have the greatest value to predict significant changes in primary and secondary endpoints at T1 and T2.

A model incorporating measures of clinical, neurophysiological and neuroimaging biomarkers could best predict individual treatment-induced behavioral gains and therefore allow to plan a "tailor-made" rehabilitation project, select rehabilitation therapy, appropriate allocation of time and human resources and stratify clinical trial enrollees.

ELIGIBILITY:
Inclusion Criteria:

* First stroke in the middle cerebral artery territory.
* Ischemic or hemorrhagic stroke (7-30 days post-acute event).
* Upper limb plegia or paresis.
* Both genders, aged >18 years.
* Ability to provide informed consent by the patient or caregiver/responsible relative.

Exclusion Criteria:

* Previous stroke.
* Stroke in territories other than the middle cerebral artery.
* Inability to provide informed consent.
* Contraindications to TMS or MRI.
* History of cancer in the past two years.
* Presence of other neurological conditions interfering with biomarkers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the Neuromotor Rehabilitation Units (Modules A-B-C) of IRCCS San Raffaele Pisana, Rome, Italy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
change in arm Fugl-Meyer score | at T0 (from 14 to 30 days post-stroke), T1 (after 2 months of intensive rehabilitation treatment) and T2 (4-6 months after discharge).
  assess the predictive power of biomarkers, individually or in combination, on the Fugl-Meyer Upper Limb Motor Scale (FM-UL) score at two months post-rehabilitation admission and at 4-6 months post-discharge

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No